CLINICAL TRIAL: NCT01613625
Title: Interest Of Renal Elastography In Children As A Diagnostic Tool Of Renal Fibrosis: Confrontation To Histological Features Of Renal Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00950-39; 2010-10 (Other: AP HM)
Record Dates: First submitted 2011-01-26; First posted 2012-06-07 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: RENAL FIBROSIS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elastography (Experimental)
  Interventions: Procedure: Elastography

INTERVENTIONS:
Procedure: Elastography

SUMMARY:
Elastography is a emerging imaging technique that has demonstrated high reliability in the assessment of tissues stiffness and quantification of fibrosis particularly in adult's livers. This ultrasound exploration has no secondary effects. There is no study published in the pediatric population concerning the role of ultrasound elastrography in kidney. The aim of this study is to look for a correlation between the elastography's results and the kidney fibrosis on children who have to undergo a renal biopsy. Elastography may play a potential diagnostic and/or prognostic role in the management of these patients which would limit invasive biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male children or feminine from 5 to 18 years old to whom is indicated a renal biopsy by the néphrologue paediatrician whatever is the initial pathology, whatever are one or several current or previous treatments and whatever is their associated comorbidity

Exclusion Criteria:

* Children of less than 5 years old or more than 18 years
* Children for whom a draining renal biopsy is not or more indicated by néphrologues
* Refusal or withdrawal of the consent lit by the holders of the exercise of the parental authority or by the child if he is capable of receiving the information
* Contraindication in the realization of a draining renal biopsy (current infection, disorder of the coagulation.)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2011-02-04 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
the elastography | 30 months
  to study a link enters the elasticity of the kidney estimated by the élastographie and the classification of the renal fibrosis estimated and quantified from the histology by draining renal biopsy.

SECONDARY OUTCOMES:
The dosage of the créatininémie | 30 months
the debit of filtration glomérulaire at the child | 30 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: alix RUOCCO, Principal Investigator — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France